CLINICAL TRIAL: NCT03481140
Title: Post-Market, Investigator Initiated, Retrospective, Audited Observational Case Series Comparing SWC With Drains to SWC With TissuGlu® and no Drains in a Donor Site DIEP Flap Breast Reconstruction Procedure in 58 Patients
Brief Title: Case Series Comparing Drains to TissuGlu® in a Donor Site DIEP Flap Breast Reconstruction Procedure
Status: Completed | Type: Observational
Sponsor: Cohera Medical, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CLN-100-0024
Record Dates: First submitted 2018-03-22; First posted 2018-03-29 (Actual); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Deep Inferior Epigastric Perforator Flap Reconstruction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Control: donor site DIEP flap breast reconstruction procedure with standard wound closure with drains
- TissuGlu Surgical Adhesive: donor site DIEP flap breast reconstruction procedure with standard wound closure with TissuGlu Surgical Adhesive and no drains
  Interventions: Device: TissuGlu Surgical Adhesive

INTERVENTIONS:
Device: TissuGlu Surgical Adhesive — lysine-derived urethane adhesive
  Groups: TissuGlu Surgical Adhesive

SUMMARY:
To evaluate the safety and effectiveness of a lysine-derived urethane adhesive (TissuGlu® Surgical Adhesive) as a less invasive alternative to surgical drains in the abdominal donor site for deep inferior epigastric perforator (DIEP) flap reconstruction.

ELIGIBILITY:
Inclusion Criteria:

* be 18 years of age or older
* be in good general health (with no conditions that would, in the opinion of the surgeon, exclude them from a drain-free donor site approach)
* have a body mass index (BMI) < 28
* have received a DIEP flap breast reconstruction procedure

Exclusion Criteria:

* current smoker
* have a body mass index (BMI) > 28
* taking active SSRI medication prescriptions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing a DIEP flap breast reconstruction at the Sana Klinik in Düsseldorf, Germany.
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2015-04-21; Primary Completion 2017-11-30 (Actual); Study Completion 2017-11-30 (Actual)

PRIMARY OUTCOMES:
number of post-operative clinical interventions related to wound fluid management at the donor site | 6 weeks post-operatively
  number of interventions

SECONDARY OUTCOMES:
total wound drainage | 6 weeks post-operatively
  drain volume + aspiration volume
cumulative drain volume | 6 weeks post-operatively
  volume
aspiration volume | 6 weeks post-operatively
  volume
cumulative days of invasive treatment | 6 weeks post-operatively
  days with drains in + days in which an aspiration was performed
days to drain removal | 6 weeks post-operatively
  days